CLINICAL TRIAL: NCT05568524
Title: The Acute and Chronic Impact of Blood Flow Restriction Resistance Training on Physical and Neuromuscular Function, Pain, and Quality of Life in Patients With Moderate/Severe Hemophilia
Brief Title: Resistance Training With Blood Flow Restriction in Hemophilia
Acronym: HemoBFR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Sofia Perez-Alenda, Dean of Faculty of Physiotherapy, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hemo-BFR-22-24
Record Dates: First submitted 2022-09-29; First posted 2022-10-05 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Hemophilia
Keywords: Hemophilia; Electromyography; Muscle Activity; Resistance Training
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): The training program for the control group consists of a telerehabilitation with traditional moderate-to-high load (60%-80% 1RM) exercises (the same as the intervention group sans BFR), utilizing elastic bands. This program for the control group will be conducted in an in-home real-time audio and video style and supervised by a physiotherapist.
  Interventions: Other: Control
- BFRT (Experimental): The BFR training program for the intervention group consists of elbow flexion and extension, and knee extension exercises performed with low load (elastic bands; equivalent to 30% 1RM) and concurrent BFR (upper limb 50% AOP; lower limb 60% AOP). Subjects will perform 4 sets (30, 15, 15 and 15 reps) of each exercise with 30 s rest between sets and 5-minute rest between exercises.
  Interventions: Other: BFRT

INTERVENTIONS:
Other: BFRT — Low-load (30% 1RM) resistance exercise with blood flow restriction
  Arms: BFRT
Other: Control — Moderate-to-high load (60%-80% 1RM) resistance exercise
  Arms: Control

SUMMARY:
The main objectives of this study are to evaluate safety and chronic effects of a low-load resistance exercise intervention (elbow flexions and extensions, and knee extensions) with blood flow restriction in people with hemophilia on quality of life, pain, and on physical and neuromuscular function.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of hemophilia A or B and undergoing prophylaxis;
* willingness to exercise twice a week during the training program and to complete the pre- and post-program evaluations;
* approval by their hematologist to participate in the exercise program;
* age between 18 and 60 years;
* informed consent signed.

Exclusion Criteria:

* the inability to attend exercise sessions at least twice a week for 8 consecutive weeks;
* non adherence to instruction on proper exercise technique;
* surgical procedures performed 6 weeks prior to or during the exercise program; - participation in any other form of exercise, not previously done, during the study;
* changes in medication during the study;
* a major bleeding episode that posed a risk or prevented exercise;
* another hemostatic defect;
* need for major surgery;
* withdrawal of informed consent.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-01-30 (Actual); Study Completion 2026-01-30 (Actual)

PRIMARY OUTCOMES:
HDsEMG | Baseline and week 8.
  Change from baseline to the end of the intervention, and the change between the intervention group and the control group.
Hand-held dynamometry (isometric elbow flexion/extension, knee extension) | Baseline and week 8.
  Change from baseline to the end of the intervention, and the change between the intervention group and the control group.
Muscle ultrasound (muscle mass, assessment of possible bleedings) | Baseline and week 8.
  Change from baseline to the end of the intervention, and the change between the intervention group and the control group.
Digital goniometry for active elbow and knee ROM | Baseline and week 8.
  Change from baseline to the end of the intervention, and the change between the intervention group and the control group.

SECONDARY OUTCOMES:
Self-reported pain intensity (Visual Analogue Scale (VAS) Scale 0-10) | Baseline and week 8.
  Change from baseline to the end of the intervention, and the change between the intervention group and the control group.
Pressure pain thresholds (digital algometry) | Baseline and week 8.
  Change from baseline to the end of the intervention, and the change between the intervention group and the control group.
Haemophilia Activities List (HAL) questionnaire | Baseline and week 8.
  The HAL measures the impact of hemophilia on self-perceived functional abilities in adults.
  Its score range is 42-252, with higher scores representing more functional limitations.
A36 haemophilia quality of life (Hemofilia-QoL) questionnaire | Baseline and week 8.
  A36 Hemofilia-QOL is a standardized disease specific questionnaire for the assessment of the health-related quality of life of people with haemophilia. The domains are physical health, daily activities, treatment satisfaction, mental aspects, relationships and social activities. There are 36 items and its score range is 0-144, with higher scores representing better outcomes.
Patient Global Impression of Change Scale (PGICS) | Baseline and week 8.
  On this scale, the patient reflects the perception of the efficacy of the treatment received in their limitation to perform activities, symptoms, emotions and overall quality of life. The PGICS consists of two subscales, one categorical and one quantitative. The categorical scale is a 7-point verbal scale with the options "I have improved a lot" = 7, "I have improved a lot" = 6, "I have improved a little" = 5, "I am the same" = 4, "I have gotten a little worse" = 3, "I have gotten a lot worse" = 2, "I have gotten a lot worse" = 1. Meanwhile, the quantitative scale consists of a line from 0 to 10, where 0 = much better and 10 = much worse.

CONTACTS AND LOCATIONS:
Overall Officials: Sofía Pérez Alenda, Principal Investigator — University of Valencia; Joaquín Calatayud, Study Chair — University of Valencia
Locations (1):
- Facultat de Fisioteràpia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No